CLINICAL TRIAL: NCT01334151
Title: A Double-blind Study of the Pharmacokinetic and Pharmacodynamic Properties of BIOD-105 and BIOD-107 Compared to Humalog® in Subjects With Type 1 Diabetes Including Assessments of Safety and Injection Site Toleration
Brief Title: Pharmacokinetic and Pharmacodynamic Properties of BIOD-105 and BIOD-107 Compared to Humalog® in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VIAject 039J
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Humalog® (Active Comparator): Humalog®, administered subcutaneously on 1 occasion
  Interventions: Drug: Insulin LISPRO
- BIOD- 105 (Experimental): BIOD- 105 administered subcutaneously on 1 occasion
  Interventions: Drug: recombinant human insulin
- BIOD-107 (Experimental): BIOD-107 administered subcutaneously on 1 occasion
  Interventions: Drug: recombinant human insulin

INTERVENTIONS:
Drug: Insulin LISPRO — Single doses of: 0.15 U/kg
  Arms: Humalog®
Drug: recombinant human insulin — Single doses of: 0.15 U/kg
  Arms: BIOD- 105; BIOD-107

SUMMARY:
The primary objective of this study is to assess the speed of absorption and onset of action of BIOD-105 and BIOD-107 and compare them to Humalog®.

DETAILED DESCRIPTION:
The secondary objectives of this study are to assess other pharmacokinetic characteristics of BIOD-105 and BIOD-107 and compare those to Humalog®, to assess other pharmacodynamic characteristics of BIOD-105 and BIOD-107 and compare those to Humalog®, and to evaluate the safety and tolerability of BIOD-105 and BIOD-107 compared to Humalog®.

ELIGIBILITY:
Inclusion Criteria:

Subjects must present with the following:

1. Body Mass Index: ≥ 18 - ≤ 28 kg/m2
2. Diagnosed with type 1 diabetes mellitus for at least 1 year
3. Insulin antibody less than or equal to 10 μU/mL at screening

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Type 2 diabetes mellitus
2. Serum C-peptide > 1.0 ng/mL
3. HbA1c > 10.0%
4. History of hypersensitivity to any of the components in the study medication
5. Treatment with any other investigational drug in the last 30 days before screening visit
6. Regular smoking as assessed clinically by the Investigator.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Speed of absorption | 480 minutes
  The speed of absorption will be assessed by the time to reach 50% of maximum insulin concentration (TINS-50%-early, time before CINS max) and the onset of action will be assessed by the time to reach 50% of the maximum glucose infusion rate (TGIR-50%- early).

CONTACTS AND LOCATIONS:
Overall Officials: Linda Morrow, MD, Principal Investigator — Profil Institute for Clinical Research, Inc. (PICR)
Locations (1):
- Profil Institute for Clinical Research, Inc. (PICR), Chula Vista, California, United States